CLINICAL TRIAL: NCT00005175
Title: Coronary Heart Disease Risk Factors in Upwardly Mobile Blacks and Whites
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1052; R29HL039788 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Hypertension; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Hypertension; Heart Diseases; Obesity

SUMMARY:
To evaluate the relation between blood pressure and socioeconomic status, electrolyte intake, obesity and psychosocial factors in Black and white students. Also, to compare blood pressure, cardiovascular risk factors, sodium and potassium excretion in United States Blacks with West African Blacks.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertension related diseases are major causes of morbidity and mortality among United States Blacks. Among Blacks and whites, lower levels of education are associated with higher levels of blood pressure, stroke, and coronary heart disease mortality. High levels of blood pressure in United States Blacks compared to United States whites persist even after controlling for education. Furthermore, it has been demonstrated that individuals living in the southeastern part of the United States continue to have higher stroke and coronary heart disease mortality rates than those living in most other areas of the United States. The number of upwardly mobile Blacks, based on education and occupation, has been increasing in the United States yet relatively little is known about the relationships of improvements in socioeconomic status and cardiovascular risk factors, particularly blood pressure. In Africa, for over four decades, hypertension has been regarded as a rare disease among the Black Africans. However, recent evidence from hospital and community based populations suggests that hypertension is the most prevalent cardiovascular disease among Africans and constitutes a major public health problem, particularly in West Africa. Furthermore, stroke is an increasing health problem.

DESIGN NARRATIVE:

In this longitudinal study, the United States students were recruited and followed annually for three years. The African students were followed for two years. At the initial clinic visit blood pressure, heart rate and anthropometric measurements were obtained and questionnaires completed concerning socioeconomic status, family and medical history, dietary practices, and smoking and drinking habits. One out of every four students had blood pressure measurements reassessed. Each participant collected an overnight urine sample for analysis of sodium and potassium. Fifty percent of the population wore a physical activity monitor for two days. Approximately ten percent of the students' families were studied to validate the hypertensive status and medical history of the parent as reported by the students and to assess known cardiovascular risk factors including obesity, smoking, alcohol intake, physical activity, and behavioral factors. Univariate analyses were conducted to assess the association between the dependent variable of blood pressure and each of the independent variables including age, body mass index, height, sodium and potassium. T-tests were used to analyze the dichotomous variables such as sex, race, and geographic location. Stratification was used to examine blood pressure levels for Blacks and whites by socioeconomic status. Multiple regression models were used to determine whether physiological or psychosocial variables were more predictive of cardiovascular risk.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1985-07; Study Completion 1990-06 (Actual)

REFERENCES:
- [Background] Adams LL, Washburn RA, Haile GT, Kuller LH. Behavioral factors and blood pressure in black college students. J Chronic Dis. 1987;40(2):131-6. doi: 10.1016/0021-9681(87)90064-6. PMID 3818866
- [Background] Washburn RA, Adams LL, Haile GT. Physical activity assessment for epidemiologic research: the utility of two simplified approaches. Prev Med. 1987 Sep;16(5):636-46. doi: 10.1016/0091-7435(87)90047-8. PMID 3684976
- [Background] Washburn RA, Adams-Campbell LL, Haile GT. Physical activity and high-density lipoprotein cholesterol and subfractions among young black adults. J Natl Med Assoc. 1987 Aug;79(8):843-8. PMID 3509873
- [Background] Adams-Campbell LL, Ukoli F, Young MP, Omene J, Nwankwo M, Haile GT, Kuller LH. An epidemiological assessment of blood pressure determinants in an adolescent population of Nigerians. J Hypertens. 1987 Oct;5(5):575-80. doi: 10.1097/00004872-198710000-00011. PMID 3429862
- [Background] Hofman A, Adams LL: Blood Pressure and Age: Is Rise of Blood Pressure During Childhood Inevitable? In: Mild Hypertension: From Drug Trials to Practice, Strasser T, Ganten D (Eds), Raven Press, New York, p 257-263, 1987
- [Background] Adams-Campbell LL, Nwankwo MU, Omene JA, Ukoli FA, Young MP, Haile GT, Kuller LH. Assessment of cardiovascular risk factors in Nigerian students. Arteriosclerosis. 1988 Nov-Dec;8(6):793-6. doi: 10.1161/01.atv.8.6.793. PMID 3196223
- [Background] Nwankwo MU, Adams-Campbell LL, Ukoli FA, Olomu IN, Ukoli CO, Ugwu E. Blood pressure in Nigerian college males. J Hum Hypertens. 1990 Apr;4(2):72-3. PMID 2338693